CLINICAL TRIAL: NCT01648751
Title: Impact of Vaginal Estrogen in the Treatment of Symptomatic Mild Pelvic Organ Prolapse With Pelvic Floor Physical Therapy
Brief Title: Vaginal Estrogen and Pelvic Floor Physical Therapy in Women With Symptomatic Mild Prolapse
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Pamela Moalli (Other)
Collaborators: American Urogynecologic Society (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Pamela Moalli, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19030408; R01HD061811 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Pelvic floor physical therapy; Vaginal estrogen; Placebo
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal estrogen (Experimental): Patients in the experimental group will receive vaginal estrogen cream
  Interventions: Drug: Vaginal estrogen
- Placebo cream (Placebo Comparator): Patients in the comparison group will receive placebo vaginal cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal estrogen — 1 gram vaginally for 7 days, followed by 1 gram vaginally twice weekly thereafter
  Other Names: Premarin vaginal cream
  Arms: Vaginal estrogen
Drug: Placebo — 1 gram vaginally for 7 days, followed by 1 gram vaginally twice weekly thereafter
  Other Names: Placebo cream
  Arms: Placebo cream

SUMMARY:
This is a randomized controlled trial in which women with symptomatic mild pelvic organ prolapse undergoing Pelvic Floor Physical Therapy (PFPT) receive vaginal estrogen versus placebo to see if a combined approach to treatment leads to improvement in clinical outcomes. The investigators predict that PFPT in combination with vaginal estrogen will lead to decreased pelvic floor symptoms and improved anatomical support corroborated by biomarker data.

DETAILED DESCRIPTION:
The pathogenesis of pelvic organ prolapse (POP) is unknown. Few studies have correlated patient symptoms and amount of prolapse with biomarkers. POP has traditionally been managed with a pessary or surgery. Recent studies suggest a reduction in POP symptoms following Pelvic Floor Physical Therapy (PFPT). Vaginally delivered hormones are also commonly used to treat prolapse symptoms, with little evidence supporting a clinical benefit. The investigators hypothesize that the optimal approach to improving prolapse symptoms in the patient with mild prolapse requires re-alignment and strengthening of levator muscles via PFPT, and optimization of tissue integrity via local estrogen therapy. The investigators propose to test this hypothesis in a randomized controlled trial in which women with symptomatic mild prolapse opting for PFPT, receive treatment with PFPT in combination with vaginal estrogen versus placebo. The investigators predict that the combined approach will lead to decreased symptoms and improved anatomical support corroborated by biomarker data.

ELIGIBILITY:
Inclusion Criteria:

* Women in good health aged 40-80
* Has symptoms of pelvic organ prolapse; answers yes to at least 1 of the following questions:

Do you feel or see a vaginal bulge? Do you feel pressure in the vagina?

* Meets POP-Q criteria on exam for stage I, II, or III prolapse
* Interested in PFPT for management of POP
* Normal mammogram within 1 year of enrollment

Exclusion Criteria:

* Prior surgery for prolapse or incontinence
* Other prior interventions for prolapse (e.g. pessary, PFPT)
* Previous bilateral salpingo-oophorectomy (women with 1 ovary will be eligible)
* Known liver dysfunction
* Connective tissue diseases known to affect collagen or elastin remodeling (including: Lupus, Rheumatoid Arthritis, Scleroderma, Sjogrens syndrome, Marfan syndrome, and Ehlers-Danlos syndrome)
* Unevaluated abnormal vaginal bleeding or abnormal pap smear in the previous year
* BMI > 35 kg/m2
* Estrogen therapy (including birth control) in the previous year
* Current or prior breast or pelvic malignancy (ovarian, tubal, uterine, cervical or vaginal)
* Contraindication to hormone use (i.e. thromboembolic disorder, use of anti-coagulants, coronary artery disease, history of stroke)

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Skoczylas, MD, MS, Study Director — University of Pittsburgh; Pamela Moalli, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was ineligible prior to randomization.
Period: Overall Study
Arm/Group | Vaginal Estrogen | Placebo Cream
Started | 9 | 11
Completed | 7 | 8
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Estrogen | Placebo Cream | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Improvement
Description: The Patient Global Impression of Improvement (PGI-I) is a global index that may be used to rate the response of a condition to a therapy (transition scale). It is a simple, direct, easy to use scale that is intuitively understandable to clinicians.
  Potential Responses:
  1. Very Much Better
  2. Much Better
  3. A Little Better
  4. No Change 5, A Little Worse
  6. Much Worse 7. Very Much Worse Lower scores indicate more imiprovment / better outcome.
Time Frame: 6 months after starting vaginal cream
Population: Subjects who completed surveys at 6 months post treatment.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Vaginal Estrogen: Patients in the experimental group will receive vaginal estrogen cream
  Vaginal estrogen: 1 gram vaginally for 7 days, followed by 1 gram vaginally twice weekly thereafter.
  The average score on the PGI-I at 6 months post treatment was 2.3. (N=7) A lower score on the PGI-I indicates improvement.
- Placebo Cream: Patients in the comparison group will receive placebo vaginal cream
  Placebo: 1 gram vaginally for 7 days, followed by 1 gram vaginally twice weekly thereafter.
  The average score on the PGI-I at 6 months post treatment was 3.0. (N=7) A lower score indicates improvement.
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 7 | 7
score on a scale | 2.3 [1 to 3] | 3.0 [1 to 5]

2. Secondary Outcome: Pelvic Floor Symptoms
Description: Pelvic Floor Symptoms, using the PFDI-20. The Pelvic Floor Distress Inventory is a condition specific quality of life instrument that assesses distress from pelvic organ prolapse, colorectal-anal, and urinary symptoms.
  Higher scores indicate greater disease burden. Range: 0 to 300
Time Frame: 6 months
Population: Subjects who completed surveys at 6 months post treatment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 7 | 7
score on a scale | 16.9 [0 to 36] | 48 [0 to 130]

3. Secondary Outcome: General Quality of Life
Description: Quality of Life, using the PFIQ-7 The Pelvic Floor Impact Questionnaire assesses how bladder, bowel, and vaginal symptoms affect activity, relationships, ad feelings.
  Higher numbers indicate greater disease burden. Score range: 0 to 300
Time Frame: 6 months
Population: Subjects who completed surveys at 6 months post treatment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 7 | 7
score on a scale | 6.1 [0 to 24] | 19.9 [0 to 76]

4. Secondary Outcome: Pelvic Organ Prolapse Stage
Description: Pelvic Organ Prolapse Stage, using the POP-Q exam. The Pelvic Organ Prolapse Quantification System use 9 measurements in the vagina to assess prolapse stage.
  Higher stage indicates greater prolapse. Range: 0 to 4
Time Frame: 6 months
Population: Subjects who underwent POP-Q measurements at 6 months post treatment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 8 | 7
units on a scale | 2 [1 to 3] | 2 [1 to 3]

5. Secondary Outcome: Collagenase Activity
Description: Collagenase Activity, via vaginal swabs collected from the posterior fornix will be used for biochemical analysis.
Time Frame: 6 months
Population: Data not available. Vaginal swabs were collected from participants. However, the lab was unable to analyze collagenase activity because there was not enough protein isolated from the samples.
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sexual Function
Description: Sexual Function, using the PISQ-12 The Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire evaluates sexual function in patients with incontinence and/or vaginal prolapse.
  Higher scores indicate greater disease burden. Scale: 0 to 48
Time Frame: 6 months
Population: Subjects who completed surveys at 6 months post treatment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Vaginal Estrogen | Placebo Cream
Number analyzed (Participants) | 7 | 6
score on a scale | 12.8 [7 to 26] | 14 [5 to 23]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vaginal Estrogen | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT01648751/Prot_SAP_000.pdf